CLINICAL TRIAL: NCT04218786
Title: Outcomes of Low-dose Colchicine in Patients With Myocardial Infarction: A Randomized Controlled Trial
Brief Title: Effect of Colchicine in Patients With Myocardial Infarction
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Due to the pandemic, there were logistical issues in continuing the study.
Sponsor: Shifa Tameer-e-Millat University (Other)
Collaborators: Rawalpindi Institute of Cardiology (Other)
Responsible Party: Principal Investigator, Nismat Javed, Principal Investigator, Shifa Tameer-e-Millat University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: STMU2020
Record Dates: First submitted 2020-01-01; First posted 2020-01-06 (Actual); Last update posted 2023-04-12 (Actual); Status verified 2023-04

CONDITIONS: Myocardium; Injury; Myocardial Infarction; Myocardial Ischemia
Keywords: colchicine; outcome: myocardial infarction
MeSH Terms: conditions — Wounds and Injuries; Myocardial Infarction; Myocardial Ischemia | interventions — Colchicine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Colchicine Group (Active Comparator): This group will receive low dose colchicine, 0.5 mg.
  Interventions: Drug: Colchicine
- Placebo group (Placebo Comparator): This group will receive a placebo drug with a similar shape and mass as that to experimental drug
  Interventions: Drug: Placebo oral tablet

INTERVENTIONS:
Drug: Colchicine — The tablet will be given once daily for the span of the study
  Arms: Colchicine Group
Drug: Placebo oral tablet — The tablet will be given once daily for the span of the study
  Arms: Placebo group

SUMMARY:
Over the past years, a substantial volume of evidence has accumulated identifying inflammatory processes as key mediators of the deleterious effects of ischemia/reperfusion-related phenomena in patients presenting with ST-segment-elevation myocardial infarction (STEMI). Nevertheless, equally impressive is the lack of clinically applicable therapeutic strategies that could mitigate these processes, thus providing significant cardioprotection. Despite the well-known fact that inflammation plays an important role in coronary artery disease development and progression, there have been few attempts to systematically examine the potential role of anti-inflammatory treatment in this setting, possibly because of a lack in anti-inflammatory agents without the adverse cardiovascular safety profile of corticosteroids and nonsteroidal anti-inflammatory drugs. Colchicine is a substance with potent anti-inflammatory properties, having a unique mechanism of action, which allows for safe use in patients with cardiovascular disease.

The purpose of the present clinical study is to test the hypothesis that a short course of treatment with colchicine could lead to reduced major adverse cardiovascular events (MACE) in acute MI.

DETAILED DESCRIPTION:
Over the past years, a substantial volume of evidence has accumulated identifying inflammatory processes as key mediators of the deleterious effects of ischemia/reperfusion-related phenomena in patients presenting with ST-segment-elevation myocardial infarction (STEMI). Nevertheless, equally impressive is the lack of clinically applicable therapeutic strategies that could mitigate these processes, thus providing significant cardioprotection.

Despite the well-known fact that inflammation plays an important role in coronary artery disease development and progression, there have been few attempts to systematically examine the potential role of anti-inflammatory treatment in this setting, possibly because of a lack in anti-inflammatory agents without the adverse cardiovascular safety profile of corticosteroids and nonsteroidal anti-inflammatory drugs. Some anti-inflammatory agents, like pexelizumab, are focused on complement cascade.Another agent is Varespladib, which targets sPLA2 that causes oxidative stress and inflammation. There are other therapeutic targets that have been widely investigated. Colchicine is a substance with potent anti-inflammatory properties, having a unique mechanism of action, which allows for safe use in patients with cardiovascular disease.

Colchicine binds to non-polymerized tubulin, forming a stable complex that effectively inhibits the dynamic of microtubules, depolymerizing them. Thus, any process requiring changes in the cell cytoskeleton, such as cellular mitosis, exocytosis and neutrophil motility, is affected. Colchicine has an important effect on atrial myocytes, changing the atrial response to autonomic effects (reducing the sympathetic activity and increasing the parasympathetic one). Due to this particular mode of action, colchicine has been indicated in atrial fibrillation post-cardiac surgery. A similar trial is being conducted to investigate any effusions or syndromes that occur after myocardial infarction.

The purpose of the present clinical study is to test the hypothesis that a short course of treatment with colchicine could lead to reduced major adverse cardiovascular events (MACE) in acute MI.

ELIGIBILITY:
Inclusion Criteria:

* All patients 18 years or above presenting in emergency department with acute myocardial infarction. These patients will be requested to take the medication at the time of discharge after stabilization and management

Exclusion Criteria:

* Patients with prior myocardial infarction 30 days before
* Patients with ischemic cardiomyopathy
* Age <18 or > 80 years
* Active inflammatory or infectious disease or known malignancy
* Known hypersensitivity to colchicine,
* renal failure (eGFR <30ml.min.1.73m)
* hepatic failure
* Stent thrombosis
* Cardiac arrest or cardiogenic shock as presenting symptoms

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2025-12 (Estimated); Primary Completion 2026-03 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Major cardiovascular adverse events (number of events) | 3 months
  This outcome will be assessed using a questionnaire. The following headings will be used:
  * Cardiovascular death (number of events)
  * Non-fatal myocardial infarction (number of events)
  * Resuscitated cardiac arrest (number of events)
  * Hospitalization for unstable angina (number of events) For each heading, the total number of events will be recorded and the numbers will all be added to calculate 'Major Adverse Cardiovascular Events' in form of number of events. This outcome has no specific values of measure but a discrete numerical value

SECONDARY OUTCOMES:
Troponin I (ng/ml) | 3 months
  This workup will be recorded on the same questionnaire as a numerical value with its specific unit of measure upon followup of patient.
Creatine Kinase-Myocardial Band (IU/L) | 3 months
  This workup will be recorded on the same questionnaire as a numerical value with its specific unit of measure upon followup of patient.
C-reactive protein (mg/L) | 3 months
  This workup will be recorded on the same questionnaire as a numerical value with its specific unit of measure upon followup of patient.

CONTACTS AND LOCATIONS:
Overall Officials: Nismat Javed, MBBS (2021), Principal Investigator — Shifa College of Medicine, Shifa Tameer-e-Millat University; Jahanzeb Malik, MBBS (2011), Study Director — Rawalpindi Institute of Cardiology; Adeel ur Rehman, MBBS, FCPS, Study Chair — Rawalpindi Institute of Cardiology
Locations (1):
- Rawalpindi Institute of Cardiology, Rawalpindi, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Turer AT, Hill JA. Pathogenesis of myocardial ischemia-reperfusion injury and rationale for therapy. Am J Cardiol. 2010 Aug 1;106(3):360-8. doi: 10.1016/j.amjcard.2010.03.032. PMID 20643246
- [Background] Christia P, Frangogiannis NG. Targeting inflammatory pathways in myocardial infarction. Eur J Clin Invest. 2013 Sep;43(9):986-95. doi: 10.1111/eci.12118. Epub 2013 Jun 17. PMID 23772948
- [Background] Adlbrecht C, Wurm R, Humenberger M, Andreas M, Redwan B, Distelmaier K, Klappacher G, Lang IM. Peri-interventional endothelin--a receptor blockade improves long-term outcome in patients with ST-elevation acute myocardial infarction. Thromb Haemost. 2014 Jul 3;112(1):176-82. doi: 10.1160/TH13-10-0832. Epub 2014 Apr 3. PMID 24695986
- [Background] He J, Li J, Wang Y, Hao P, Hua Q. Neutrophil-to-lymphocyte ratio (NLR) predicts mortality and adverse-outcomes after ST-segment elevation myocardial infarction in Chinese people. Int J Clin Exp Pathol. 2014 Jun 15;7(7):4045-56. eCollection 2014. PMID 25120783
- [Background] Kawaguchi M, Takahashi M, Hata T, Kashima Y, Usui F, Morimoto H, Izawa A, Takahashi Y, Masumoto J, Koyama J, Hongo M, Noda T, Nakayama J, Sagara J, Taniguchi S, Ikeda U. Inflammasome activation of cardiac fibroblasts is essential for myocardial ischemia/reperfusion injury. Circulation. 2011 Feb 15;123(6):594-604. doi: 10.1161/CIRCULATIONAHA.110.982777. Epub 2011 Jan 31. PMID 21282498
- [Background] Chen K, Schenone AL, Borges N, Militello M, Menon V. Teaching an Old Dog New Tricks: Colchicine in Cardiovascular Medicine. Am J Cardiovasc Drugs. 2017 Oct;17(5):347-360. doi: 10.1007/s40256-017-0226-3. PMID 28353024
- [Background] Robertson S, Martinez GJ, Payet CA, Barraclough JY, Celermajer DS, Bursill C, Patel S. Colchicine therapy in acute coronary syndrome patients acts on caspase-1 to suppress NLRP3 inflammasome monocyte activation. Clin Sci (Lond). 2016 Jul 1;130(14):1237-46. doi: 10.1042/CS20160090. Epub 2016 Apr 21. PMID 27129183
- [Background] Misawa T, Takahama M, Kozaki T, Lee H, Zou J, Saitoh T, Akira S. Microtubule-driven spatial arrangement of mitochondria promotes activation of the NLRP3 inflammasome. Nat Immunol. 2013 May;14(5):454-60. doi: 10.1038/ni.2550. Epub 2013 Mar 17. PMID 23502856
- [Background] Akodad M, Fauconnier J, Sicard P, Huet F, Blandel F, Bourret A, de Santa Barbara P, Aguilhon S, LeGall M, Hugon G, Lacampagne A, Roubille F. Interest of colchicine in the treatment of acute myocardial infarct responsible for heart failure in a mouse model. Int J Cardiol. 2017 Aug 1;240:347-353. doi: 10.1016/j.ijcard.2017.03.126. Epub 2017 Apr 1. PMID 28395979
- [Background] Rymer JA, Newby LK. Failure to Launch: Targeting Inflammation in Acute Coronary Syndromes. JACC Basic Transl Sci. 2017 Aug 28;2(4):484-497. doi: 10.1016/j.jacbts.2017.07.001. eCollection 2017 Aug. PMID 30062164
- [Background] Pinckard RN, Olson MS, Giclas PC, Terry R, Boyer JT, O'Rourke RA. Consumption of classical complement components by heart subcellular membranes in vitro and in patients after acute myocardial infarction. J Clin Invest. 1975 Sep;56(3):740-50. doi: 10.1172/JCI108145. PMID 808560
- [Background] Gora S, Maouche S, Atout R, Wanherdrick K, Lambeau G, Cambien F, Ninio E, Karabina SA. Phospholipolyzed LDL induces an inflammatory response in endothelial cells through endoplasmic reticulum stress signaling. FASEB J. 2010 Sep;24(9):3284-97. doi: 10.1096/fj.09-146852. Epub 2010 Apr 29. PMID 20430794
- [Background] Serruys PW, Garcia-Garcia HM, Buszman P, Erne P, Verheye S, Aschermann M, Duckers H, Bleie O, Dudek D, Botker HE, von Birgelen C, D'Amico D, Hutchinson T, Zambanini A, Mastik F, van Es GA, van der Steen AF, Vince DG, Ganz P, Hamm CW, Wijns W, Zalewski A; Integrated Biomarker and Imaging Study-2 Investigators. Effects of the direct lipoprotein-associated phospholipase A(2) inhibitor darapladib on human coronary atherosclerotic plaque. Circulation. 2008 Sep 9;118(11):1172-82. doi: 10.1161/CIRCULATIONAHA.108.771899. Epub 2008 Sep 1. PMID 18765397
- [Background] Ridker PM, Thuren T, Zalewski A, Libby P. Interleukin-1beta inhibition and the prevention of recurrent cardiovascular events: rationale and design of the Canakinumab Anti-inflammatory Thrombosis Outcomes Study (CANTOS). Am Heart J. 2011 Oct;162(4):597-605. doi: 10.1016/j.ahj.2011.06.012. Epub 2011 Sep 14. PMID 21982649
- [Background] Tanguay JF, Geoffroy P, Sirois MG, Libersan D, Kumar A, Schaub RG, Merhi Y. Prevention of in-stent restenosis via reduction of thrombo-inflammatory reactions with recombinant P-selectin glycoprotein ligand-1. Thromb Haemost. 2004 Jun;91(6):1186-93. doi: 10.1160/TH03-11-0701. PMID 15175806
- [Background] Surinkaew S, Kumphune S, Chattipakorn S, Chattipakorn N. Inhibition of p38 MAPK during ischemia, but not reperfusion, effectively attenuates fatal arrhythmia in ischemia/reperfusion heart. J Cardiovasc Pharmacol. 2013 Feb;61(2):133-41. doi: 10.1097/FJC.0b013e318279b7b1. PMID 23107875
- [Background] Fujisue K, Sugamura K, Kurokawa H, Matsubara J, Ishii M, Izumiya Y, Kaikita K, Sugiyama S. Colchicine Improves Survival, Left Ventricular Remodeling, and Chronic Cardiac Function After Acute Myocardial Infarction. Circ J. 2017 Jul 25;81(8):1174-1182. doi: 10.1253/circj.CJ-16-0949. Epub 2017 Apr 18. PMID 28420825
- [Background] Martinez GJ, Robertson S, Barraclough J, Xia Q, Mallat Z, Bursill C, Celermajer DS, Patel S. Colchicine Acutely Suppresses Local Cardiac Production of Inflammatory Cytokines in Patients With an Acute Coronary Syndrome. J Am Heart Assoc. 2015 Aug 24;4(8):e002128. doi: 10.1161/JAHA.115.002128. PMID 26304941
- [Background] Deftereos S, Giannopoulos G, Angelidis C, Alexopoulos N, Filippatos G, Papoutsidakis N, Sianos G, Goudevenos J, Alexopoulos D, Pyrgakis V, Cleman MW, Manolis AS, Tousoulis D, Lekakis J. Anti-Inflammatory Treatment With Colchicine in Acute Myocardial Infarction: A Pilot Study. Circulation. 2015 Oct 13;132(15):1395-403. doi: 10.1161/CIRCULATIONAHA.115.017611. Epub 2015 Aug 11. PMID 26265659
- [Background] Singhal R, Chang SL, Chong E, Hsiao YW, Liu SH, Tsai YN, Hsu CP, Lin YJ, Lo LW, Ha TL, Chen YC, Chen YJ, Chiou CW, Chen SA. Colchicine suppresses atrial fibrillation in failing heart. Int J Cardiol. 2014 Oct 20;176(3):651-60. doi: 10.1016/j.ijcard.2014.07.069. Epub 2014 Aug 17. PMID 25164186
- [Background] Imazio M, Brucato A, Cemin R, Ferrua S, Maggiolini S, Beqaraj F, Demarie D, Forno D, Ferro S, Maestroni S, Belli R, Trinchero R, Spodick DH, Adler Y; ICAP Investigators. A randomized trial of colchicine for acute pericarditis. N Engl J Med. 2013 Oct 17;369(16):1522-8. doi: 10.1056/NEJMoa1208536. Epub 2013 Aug 31. PMID 23992557
- [Background] Tardif JC, Kouz S, Waters DD, Bertrand OF, Diaz R, Maggioni AP, Pinto FJ, Ibrahim R, Gamra H, Kiwan GS, Berry C, Lopez-Sendon J, Ostadal P, Koenig W, Angoulvant D, Gregoire JC, Lavoie MA, Dube MP, Rhainds D, Provencher M, Blondeau L, Orfanos A, L'Allier PL, Guertin MC, Roubille F. Efficacy and Safety of Low-Dose Colchicine after Myocardial Infarction. N Engl J Med. 2019 Dec 26;381(26):2497-2505. doi: 10.1056/NEJMoa1912388. Epub 2019 Nov 16. PMID 31733140
- [Background] Deftereos S, Giannopoulos G, Papoutsidakis N, Panagopoulou V, Kossyvakis C, Raisakis K, Cleman MW, Stefanadis C. Colchicine and the heart: pushing the envelope. J Am Coll Cardiol. 2013 Nov 12;62(20):1817-25. doi: 10.1016/j.jacc.2013.08.726. Epub 2013 Sep 11. PMID 24036026
- [Background] Head BP, Patel HH, Roth DM, Murray F, Swaney JS, Niesman IR, Farquhar MG, Insel PA. Microtubules and actin microfilaments regulate lipid raft/caveolae localization of adenylyl cyclase signaling components. J Biol Chem. 2006 Sep 8;281(36):26391-9. doi: 10.1074/jbc.M602577200. Epub 2006 Jul 3. PMID 16818493
- [Background] Malan D, Gallo MP, Bedendi I, Biasin C, Levi RC, Alloatti G. Microtubules mobility affects the modulation of L-type I(Ca) by muscarinic and beta-adrenergic agonists in guinea-pig cardiac myocytes. J Mol Cell Cardiol. 2003 Feb;35(2):195-206. doi: 10.1016/s0022-2828(02)00312-7. PMID 12606260
- [Background] Imazio M, Brucato A, Ferrazzi P, Rovere ME, Gandino A, Cemin R, Ferrua S, Belli R, Maestroni S, Simon C, Zingarelli E, Barosi A, Sansone F, Patrini D, Vitali E, Trinchero R, Spodick DH, Adler Y; COPPS Investigators. Colchicine reduces postoperative atrial fibrillation: results of the Colchicine for the Prevention of the Postpericardiotomy Syndrome (COPPS) atrial fibrillation substudy. Circulation. 2011 Nov 22;124(21):2290-5. doi: 10.1161/CIRCULATIONAHA.111.026153. Epub 2011 Nov 16. PMID 22090167
- [Background] Zarpelon CS, Netto MC, Jorge JC, Fabris CC, Desengrini D, Jardim Mda S, Silva DG. Colchicine to Reduce Atrial Fibrillation in the Postoperative Period of Myocardial Revascularization. Arq Bras Cardiol. 2016 Jul;107(1):4-9. doi: 10.5935/abc.20160082. Epub 2016 May 24. PMID 27223641
- [Background] Imazio M, Belli R, Brucato A, Ferrazzi P, Patrini D, Martinelli L, Polizzi V, Cemin R, Leggieri A, Caforio AL, Finkelstein Y, Hoit B, Maisch B, Mayosi BM, Oh JK, Ristic AD, Seferovic P, Spodick DH, Adler Y. Rationale and design of the COlchicine for Prevention of the Post-pericardiotomy Syndrome and Post-operative Atrial Fibrillation (COPPS-2 trial): a randomized, placebo-controlled, multicenter study on the use of colchicine for the primary prevention of the postpericardiotomy syndrome, postoperative effusions, and postoperative atrial fibrillation. Am Heart J. 2013 Jul;166(1):13-9. doi: 10.1016/j.ahj.2013.03.025. Epub 2013 May 6. PMID 23816016
- [Background] Imazio M, Bobbio M, Cecchi E, Demarie D, Demichelis B, Pomari F, Moratti M, Gaschino G, Giammaria M, Ghisio A, Belli R, Trinchero R. Colchicine in addition to conventional therapy for acute pericarditis: results of the COlchicine for acute PEricarditis (COPE) trial. Circulation. 2005 Sep 27;112(13):2012-6. doi: 10.1161/CIRCULATIONAHA.105.542738. PMID 16186437
- [Background] Imazio M, Bobbio M, Cecchi E, Demarie D, Pomari F, Moratti M, Ghisio A, Belli R, Trinchero R. Colchicine as first-choice therapy for recurrent pericarditis: results of the CORE (COlchicine for REcurrent pericarditis) trial. Arch Intern Med. 2005 Sep 26;165(17):1987-91. doi: 10.1001/archinte.165.17.1987. PMID 16186468
- [Background] Imazio M, Brucato A, Cemin R, Ferrua S, Belli R, Maestroni S, Trinchero R, Spodick DH, Adler Y; CORP (COlchicine for Recurrent Pericarditis) Investigators. Colchicine for recurrent pericarditis (CORP): a randomized trial. Ann Intern Med. 2011 Oct 4;155(7):409-14. doi: 10.7326/0003-4819-155-7-201110040-00359. Epub 2011 Aug 28. PMID 21873705
- [Background] Imazio M, Belli R, Brucato A, Cemin R, Ferrua S, Beqaraj F, Demarie D, Ferro S, Forno D, Maestroni S, Cumetti D, Varbella F, Trinchero R, Spodick DH, Adler Y. Efficacy and safety of colchicine for treatment of multiple recurrences of pericarditis (CORP-2): a multicentre, double-blind, placebo-controlled, randomised trial. Lancet. 2014 Jun 28;383(9936):2232-7. doi: 10.1016/S0140-6736(13)62709-9. Epub 2014 Mar 30. PMID 24694983
- [Background] Verma S, Eikelboom JW, Nidorf SM, Al-Omran M, Gupta N, Teoh H, Friedrich JO. Colchicine in cardiac disease: a systematic review and meta-analysis of randomized controlled trials. BMC Cardiovasc Disord. 2015 Aug 29;15:96. doi: 10.1186/s12872-015-0068-3. PMID 26318871
- [Background] Leung YY, Yao Hui LL, Kraus VB. Colchicine--Update on mechanisms of action and therapeutic uses. Semin Arthritis Rheum. 2015 Dec;45(3):341-50. doi: 10.1016/j.semarthrit.2015.06.013. Epub 2015 Jun 26. PMID 26228647
- [Background] Terkeltaub RA, Furst DE, Digiacinto JL, Kook KA, Davis MW. Novel evidence-based colchicine dose-reduction algorithm to predict and prevent colchicine toxicity in the presence of cytochrome P450 3A4/P-glycoprotein inhibitors. Arthritis Rheum. 2011 Aug;63(8):2226-37. doi: 10.1002/art.30389. PMID 21480191